CLINICAL TRIAL: NCT02391740
Title: THERAPEUTIC PATIENT EDUCATION AND CANCER PAIN
Acronym: EFFADOL
Status: Completed | Type: Observational
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-A00239-38
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Questionnaire

SUMMARY:
Describe the expectations of therapeutic education for patients in management of cancer pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient with cancer diagnosed for at least one month
* Patient with pain from the tumor or its treatment
* Patients with a life expectancy ≥ 6 months
* Health condition compatible with the requirements of the program (WHO performance scale < or= 2)
* Age over 18 years
* Patient able to understand, speak and read French
* Absence of cognitive impairment

Exclusion Criteria:

* Primary cancer of the central nervous system or brain metastases
* Disorders of the documented higher functions
* Evolutionary psychiatric pathology
* Drug User
* Abusive alcohol consumption than the WHO recommendations (or 3 glasses of wine per day)
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cancer and pain
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2015-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
describe the expectations of therapeutic education for patients in management of cancer pain | at inclusion

SECONDARY OUTCOMES:
Describe the expectations of close person in therapeutic education on management of cancer pain | at inclusion
Estimate the intensity of the pain | at inclusion
Estimate the echo of the pain on the daily activity of the patient | at inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- centre François Baclesse, Caen, France